CLINICAL TRIAL: NCT04089254
Title: A Multi-Site Study to Compare the Outcomes of Psychiatric Treatment of Suicidal Adolescents in Different Treatment Settings
Brief Title: Suicide Treatment Alternatives for Teens
Acronym: START
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS-2018C1-11111
Record Dates: First submitted 2019-07-09; First posted 2019-09-13 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Suicidal Ideation
Keywords: Suicide; Suicidal; Adolescent
MeSH Terms: conditions — Suicidal Ideation; Suicide

STUDY DESIGN:
Intervention Model Description: Quasi-Randomized Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient Psychiatry (Active Comparator): Child and adolescent inpatient treatment
  Interventions: Behavioral: Inpatient Psychiatry
- Outpatient Crisis Intervention Clinic (Active Comparator): OCIC is outpatient crisis intervention clinic
  Interventions: Behavioral: Outpatient Crisis Intervention Clinic

INTERVENTIONS:
Behavioral: Inpatient Psychiatry — Inpatient hospitalization to treat and stabilize suicidal thoughts and behavior.
  Arms: Inpatient Psychiatry
Behavioral: Outpatient Crisis Intervention Clinic — Outpatient psychiatric clinic that provides crisis intervention to treat and stabilize suicidal thoughts and behavior.
  Arms: Outpatient Crisis Intervention Clinic

SUMMARY:
Quasi-Randomized trial to compare inpatient care versus outpatient crisis intervention clinic. This study plans to enroll up to 1,000 participants across 4 sites in a 5 years period.

DETAILED DESCRIPTION:
To address the unmet need of optimizing the treatment and management for adolescent suicidality, the investigators propose to evaluate if Outpatient Crisis Intervention Clinic (OCIC) leads to better treatment outcomes than inpatient treatment. To achieve this goal, the investigators propose a multi- site study to evaluate if OCIC, compared with inpatient care, can lead to a lower risk of a suicidal event (primary outcome) as well as higher treatment satisfaction (TS) and satisfaction with life (SL) (secondary outcomes) of both the legal guardians/parents and patients. Furthermore, the investigators will assess which clinical and socioeconomic factors at baseline may affect the treatment outcomes. With the results from the proposed study, the investigators will be able to reduce the family and clinician decisional uncertainty about the best treatment setting for suicidal adolescents in the target population. The results will significantly help patients, families, and clinicians with this decision-making process and improve outcomes for suicidal adolescents. The study has been designed to accomplish the following Specific Aims (SA):

SA1: Measure the differences between OCIC and inpatient treatment in the time to first recurrence of a suicidal event (a suicide attempt, interrupted attempt, hospitalization because of suicidal risk, an emergency/urgent evaluation because of suicidal risk, and a death by suicide) and the number of suicidal events over 30 days, 90 days and 180 days for suicidal adolescents after their baseline Emergency Department (ED) visits.

Hypothesis (H) 1.1: Assignment with randomization to OCIC from the ED will lead to a longer time to the first recurrence of a suicidal event compared to inpatient treatment after 30 days, 90 days and 180 days from the baseline ED visit for suicidality. H1.2 Assignment with randomization to OCIC will lead to a lower number suicidal events over 30 days, 90 days and 180 days when compared to inpatient treatment. H1.3 Heterogeneity of Treatment Effects [HTE]: The investigators will examine to what degree the following specific clinical features and sociodemographic features differ for patients who respond to OCIC or inpatient psychiatry treatment. Response is defined by a delay in first recurrence of a suicidal event and a lower number of suicidal events over 30 days, 90 days and 180 days. Clinical features: 1) Severity of suicidal ideation at baseline and over 180 days; 2) number of suicidal events at baseline only; 3) Substance use at baseline and over 180 days. Sociodemographic features at baseline: 1) Age 2) Gender 3) Gender Identity 4) Type of Insurance (public insurance/no insurance/private) 5) Ethnicity (Hispanic/Non); 6) Race (African-American (AA) versus non-African American); 7) Living with one biological parent, two biological parents, a stepparent, a relative, or other SA2: Assess the treatment satisfaction (TS) and satisfaction with life (SL) across OCIC and inpatient treatment.

H2.1: Overall, patients and legal guardians/parents in the OCIC group will have higher TS (at the completion of treatment in OCIC or inpatient psychiatry) and better SL than the inpatient treatment group over30 days, 90 and 180 days.

SA3: As an exploratory aim, assess the demographics and potential barriers to treatment for a third comparator of the "no show" group who were randomized to OCIC or inpatient treatment but never showed up or left the inpatient unit against medical advice (AMA).

H3.1: The no show group (the third comparator) who did not arrive for any OCIC appointments or left AMA from inpatient treatment will differ from the other comparators with respect to the following barriers to treatment: 1) Age 2) Gender 3) Type of Insurance (public insurance/no insurance/private) 4) Ethnicity (Hispanic/Non) 64; 5) Race (African-American (AA) versus non-African American) ; 6) Living with one biological parent, two biological parents, a stepparent, a relative, or other H3.2: The no show group will have significantly shorter time to first recurrence of a suicidal event and a larger number of suicidal events over 30 days, 90 days and 180 days in comparison to the other patients.

SA4: As a secondary aim, evaluate the difference of outcomes (see outcomes in SA1 and SA2) in week-by-week treatment allocation followers and treatment switchers.

SA 5: As a secondary aim, evaluate the difference in outcomes between in-person OCIC services and telehealth OCIC services.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents that are 12 through 17 years old (including 17 year olds who will turn 18 years old during the course of the study).
2. Are brought to the Emergency Department (ED) due to suicidal thoughts or behaviors
3. Require a higher level of care (OCIC or Inpatient) indicated by clinician determination and a CHRT-SR score of 15 to 52.
4. The presence of a legal guardian
5. Capable of giving signed informed consent/assent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Adolescents with suicidal thoughts that place themselves at a serious imminent risk of suicide based on clinical judgment.
2. Adolescents who require 24 hour/day supervision but no adult can provide 24 hour/day supervision outside of the hospital
3. Adolescents without the ability to read and answer survey questions
4. Adolescents that are non-English speaking due to the scales and surveys that are used for this study only being available in English.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Time to first recurrence of a suicide event | 180 days
  Measure the differences between OCIC and inpatient treatment in the time to first recurrence of a suicidal event (a suicide attempt, interrupted attempt, hospitalization because of suicidal risk, an emergency/urgent evaluation because of suicidal risk, and a death by suicide).
Number of suicide events after treatment. | 180 days
  Measure the difference between OCIC and inpatient treatment in the number of suicidal events (a suicide attempt, interrupted attempt, hospitalization because of suicidal risk, an emergency/urgent evaluation because of suicidal risk, and a death by suicide) over 180 days for suicidal adolescents after their baseline ED visit.

SECONDARY OUTCOMES:
Treatment Satisfaction as assessed using the Client Satisfaction Questionnaire-Adapted (CSQ). | 180 days
  Assess the rate of client treatment satisfaction (TS) across OCIC and inpatient treatment. This will be measured by patient completing the Client Satisfaction Questionnaire-Adapted (CSQ).
Demographic factors as assessed using the START demographics form. | 180 days
  As an exploratory aim, assess the demographic influences that may impact treatment outcomes for all groups (inpatient, OCIC, and no show group).This will be measured by the patient and parent completing the START demographics form, including information on race, ethnicity, patient sexual orientation, patient sexual identify, household education level and income, family makeup (number of parents and/or guardians in the home), and other socio-economic factors.
Quality of Life Satisfaction as assessed using the PROMIS® (Patient-Reported Outcomes Measurement Information System) Item Bank v1.0 - General Life Satisfaction - Short Form 5a | 180 days
  Assess and compare the patient's life satisfaction following treatment in either OCIC or inpatient using the PROMIS® (Patient-Reported Outcomes Measurement Information System) Item Bank v1.0 - General Life Satisfaction - Short Form 5a.
Quality of Life Satisfaction as assessed using the PROMIS Pediatric Item Bank v1.0 - Life Satisfaction - Short Form 4a | 180 days
  Assess and compare the patient's life satisfaction following treatment in either OCIC or inpatient using the Quality of Life Satisfaction as assessed using the PROMIS Pediatric Item Bank v1.0 - Life Satisfaction - Short Form 4a.
Quality of Life Satisfaction as assessed using PROMIS Parent Proxy Item Bank v1.0 - Life Satisfaction - Short Form 8a | 180 days
  Assess and compare the patient's life satisfaction following treatment in either OCIC or inpatient using the : Quality of Life Satisfaction as assessed using PROMIS Parent Proxy Item Bank v1.0 - Life Satisfaction - Short Form 8a.

CONTACTS AND LOCATIONS:
Overall Officials: Drew Barzman, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Northwell Health, Glen Oaks, New York
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - UT Southwestern Medical Center/Children's Health, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CDC, Web-based Injury Statistics Query and Reporting System — http://www.cdc.gov/injury/wisqars/index.html